CLINICAL TRIAL: NCT01566487
Title: Randomized, Open-Label, Balanced, Two-treatment, Two-period, Two-sequence, Crossover, Multicentric Experimental Bioequivalence Study of Quetiapine Fumarate Film-coated Tablets 300 mg (Test)and Seroquel Film-coated Tablets 300 mg (Reference) Under Fasting Condition
Brief Title: Bioequivalence Study of Quetiapine Fumarate Tablets 300 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 353-09
Record Dates: First submitted 2012-03-28; First posted 2012-03-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
Keywords: Bioequivalence; Quetiapine fumarate; crossover
MeSH Terms: interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine fumarate tablets 300 mg (Experimental): Quetiapine fumarate film-coated tablets 300 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Quetiapine fumarate
- Seroquel (Active Comparator): Seroquel film-coated tablets 300 mg of Astrazeneca Pharmaceuticals, USA
  Interventions: Drug: Quetiapine fumarate

INTERVENTIONS:
Drug: Quetiapine fumarate — Quetiapine fumarate tablets 300mg
  Other Names: Seroquel

SUMMARY:
This is an open label, randomised, balanced, two-treatment, two-period, two-sequence, crossover, multicentric experimental bioequivalence study.

DETAILED DESCRIPTION:
The objective of this study was to compare the bioavailability and characterise the pharmacokinetics profile of the sponsor formulation Quetiapine fumarate tablets 300 mg of Dr. Reddy's Laboratories Limited, India with respect to reference formulation Seroquel tablets 300 mg of Astrazeneca Pharmaceuticals, USA in adults schizophrenia patients under fasting condition.

54 subjects were dosed and were enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for participation in the study by the patient and Patient's Legally Acceptable Representative (LAR). If the patient or his/her legally acceptable representative is unable to read/write - an impartial witness should be present during the entire informed consent process who must append his/her signatures to the consent form.
* Schizophrenic patients, between 18 and 55 years of age (inclusive).
* Patient has a documented clinical diagnosis of stable schizophrenia (DSM IV-TR) controlled by a stable 300 mg Quetiapine regimen given at 12-hour intervals from at least 2 weeks prior to the first dosing, as confirmed by Principal Investigator
* Having a Body Mass Index (BMI) between 18 and 35 (inclusive). calculated as weight in kg/height in m2.
* Not having any significant diseases or clinically significant abnormal findings except schizophrenia during screening, medical history, physical examination, laboratory evaluations, 12-lead ECG recordings and Chest X ray (Postero-anterior view).
* The investigator must ensure that the respective hepatic, renal, haematopoietic, cardiac and respiratory functions are appropriate to include the patient in the study.
* Able to comply with study procedures in the opinion of the investigator.
* In case of female patient the serum pregnancy test at screening visit must be negative.
* Sexually active women, unless surgically sterile (at least 6 months prior to Study drug administration) or postmenopausal for at least 12 consecutive months, must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives [any hormonal method in conjunction with a secondary method], intrauterine device, female condom with spermicide. diaphragm with spermicide.Absolute sexual abstinence, use of condom with spermicide by sexual partner or sterile [at least 6 months prior to Study drug administration] sexual partner) for at least 4 weeks prior to study drug administration,during study and up to 30 days after the last dose of study drug. Cessation of birth control after this point should be discussed with a responsible physician. (It is investigator's responsibility to ensure that above points regarding an effective method of avoiding pregnancy are discussed with patient/LAR in detail and patient agreed for this and it is documented in source document. The investigator should ensure that the patient is using an effective method of avoiding pregnancy as per protocol).
* In case of Male patients: Either partner or patient must use an effective method of avoiding pregnancy for at least 4 weeks prior to study drug administration, during study and up to 30 days after the last dose of study drug. Cessation of birth control after this point should be discussed with a responsible physician.
* (It is investigator's responsibility to ensure that above points regarding an effective method of avoiding pregnancy are discussed with patient/LAR in detail and patient agreed for this and it is documented in source document. The investigator should ensure that the patient is using an effective method of avoiding pregnancy as per protocol).

Exclusion Criteria:

* Known hypersensitivity/allergy or idiosyncratic reaction to Quetiapine or its excipients.
* Clinically significant illnesses (including hypotensive episodes and systemic infection) or surgery within 4 weeks prior to the first dosing.
* Current or relevant history of serious. severe or unstable psychiatric illness (Meeting the criteria for any other (Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) AXIS I) except schizophrenia.
* History of syncope or orthostatic hypotension
* Ingestion of any medication other than listed below at any time in 10 days before the first study drug administration. In any such case Patient selection will be at the discretion of the Principal Investigator.

Following is the list of permissible medications, provided, the patients are on a stable regimen at least I0 days prior to and throughout the study.

Alprazolam, Fluoxetin, Imipramine, Haloperidol, Risperidone. (Refer Appendix 4 for list of nonpermissible medication)

* A history of alcohol or drug dependence by DSM-IV criteria within 6 months prior to screening.
* Smokers who smoke 10 or more than 10 cigarette/day or inability to abstain from smoking during the study
* Donation of blood (≥ 1 unit or 350 mL) within 90 days prior to receiving the first dose of study medication or during the study.

Note: In case the blood loss is less than or equol to 200 mL; patient may be dosed 60 days after blood donation.

* A positive hepatitis screen including hepatitis B surface antigen or HCV antibodies.
* Positive test for HIV infection.
* ECG abnormalities (clinically relevant), vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mnHg, diastolic blood pressure lower than 50 or over 90 mmHg or patient on any antihypertensive medication or heart rate less than 50 or over 100 bpm) or significant orthostatic hypotension (i.e.. a drop in systolic blood pressure of 30 mmHg or more and/or a drop in diastolic blood pressure of 20 mmHg or more on standing) at screening. Patients with vital signs values no more than 5% out of the specified range but considered stable could be included in the study at the discretion of the investigator.
* Any condition1 Abnormal baseline findings that in the investigator's judgement might increase the risk to the patient or decrease the chance of obtaining satisfactory data needed to obtain the objective of the study.
* The receipt of an investigational product or participation in a drug research study within a period of 30 days prior to the first dose of study medication.

Note: Elimination half-life of the study drug should be taken into consideration for inclusion of the Patient in the study.

* Psychosis judged to be the direct physiological effect of an abused medication or substance.
* Positive testing for the drugs of abuse (amphetamines, barbiturates ,benzodiazepines, cocaine, morphine, marijuana) done by urine scan at Screening. (Except for alprazolam which is a permissible medication).
* Known history of Organic Brain Disorder.
* Hospitalisation for an exacerbation of schizophrenia within two months prior to screening and during the screening period.
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Patients with the following cardiac conditions are excluded:

  * Recent myocardial infarction (<I2 months)
  * QTc prolongation (screening electrocardiogram with QTc > 450 msec for men, QTc > 470 msec for women)
* History of QTc prolongation or using concomitant medications which prolong QTc interval

  * Sustained cardiac arrhythmia or history of sustained cardiac arrhythmia
  * Uncompensated congestive heart failure
  * Complete left bundle branch block
  * First-degree heart block with PR interval > 0.22 seconds
* Presence of cataract on Ophthalmoscopic examination (slit lamp exam).
* History of agranulocytosis.
* Known case of Diabetes mellitus or fasting blood glucose ≥126 mg/dl at screening visit.
* Clinically significant history or presence of any gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease (e.g, hepatic insufficiency), or other conditions known to interfere with the absorption, distribution,metabolism, or excretion of the drug.
* Concurrent Parkinson's disease
* Clinically significant history of cataracts, tardive dyskinesia. neuroleptics malignant syndrome. epilepsy or seizure.
* Any clinically relevant neurological, endocrinal. cardiovascular. cerebrovascular, pulmonary, hematological, or immunologic disease could lead to safety risk to the patient upon participation in the trial or could interfere with the conduct of the trial
* Any reason that, in the opinion of the Investigator, would prevent the patient from participating in the study.
* Patients with abnormal thyroid function test at screening visit which as judged by Investigator could lead to safety risk to the patient upon participation in the trial or could Interfere with the conduct of the trial.
* Patient with hyperprolactinemia at screening visit which as judged by Investigator could lead to safety risk to the patient upon participation in the trial or could interfere with the conduct of the trial.
* Dementia related psychosis.
* Pregnant or lactating females

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Area under curve(AUC) | Period 1 - Pre-dose in day 3, 4 and 5 and period 2 pre dose in day8,9 and 10 and 0.25,0.5,0.75,1.25,1.5,1.75,2,2.5,3,4,6,8,10 & 12 hrs post-dose on day 5 and day 10

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Sachin Patkar, MD, Principal Investigator — Masina hospital
Locations (1):
- Lambda Therapeutic Research Ltd, Ahmedabad, Gujarat, India